CLINICAL TRIAL: NCT01544452
Title: Prospective Randomized Study of Total Preoperative MR Diagnostic Evaluation Versus Standard Diagnostic Evaluation in Patients With Rectal Cancer
Brief Title: Total Preoperative MR Diagnostic Evaluation Versus Standard Diagnostic Evaluation in Patients With Rectal Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of MR scanning capacity
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Michael Achiam, Senior Resident, M.D., ph.d., Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: H-1-2009-094
Record Dates: First submitted 2011-11-07; First posted 2012-03-06 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Rectal Cancer; Liver Metastasis
Keywords: MR; CT; ultrasonography; MR colonography; MR rectum; MR liver
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Total preoperative MR evaluation (Other): Total diagnostic evaluation with MRI of the liver, abdomen, colonography and rectum in one session combined with CT thorax
  Interventions: Procedure: MR colonography and MR of the liver
- Standard diagnostic evaluation (Other): Standard preoperative diagnostic evaluation for patients with rectal cancer, incl. CT thorax, abdomen and MRI of the rectum and colonoscopy
  Interventions: Procedure: Standard diagnostic evaluation

INTERVENTIONS:
Procedure: MR colonography and MR of the liver — Altered planned surgical procedure if MR colonoscopy reveals synchronous cancer or larger polyps
  Other Names: Total preoperative MR evaluation
  Arms: Total preoperative MR evaluation
Procedure: Standard diagnostic evaluation — Altered planned surgical procedure if MR colonoscopy reveals synchronous cancer or larger polyps
  Arms: Standard diagnostic evaluation

SUMMARY:
Patients with rectal cancer undergo MRI of the rectum, CT of the thorax and abdomen (or thorax x-ray and ultrasonic liver evaluation) and colonoscopy as a total diagnostic evaluation before surgery. MR colonography have been shown to have high sensitivity and specificity for larger polyps and cancer and MRI of the liver have been shown to have similar or higher sensitivity than CT of the liver for metastasis. Since patients already undergo MR of the rectum, the investigators have proposed a total diagnostic evaluation with MRI of the liver, abdomen, colonography and rectum in one session (minus thorax evaluation) instead of two or three different methods of evaluation. The investigators hypothesis is that the total MR evaluation is equal or superior to the existing preoperative evaluation regarding the diagnosis of synchronous cancers and liver metastasis and regarding cost-benefit for the total diagnostic evaluation.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is among the most common cancer forms in Denmark with an approximate of 4300 new cases in Denmark annually, of which rectal cancer represents approximately 1400 new cases each year. It is also well known that synchronous cancer and polyps are present in up to 11% and 58% respectively in patients with CRC. It is assumed that adenomas constitute a precursor for cancer and it is thus speculated that the detection and removal of the adenoma could reduce the incidence and mortality of colorectal cancer. Danish Colorectal Cancer Group (DCCG) and the Danish Surgical Society (DKS) currently recommend full colonic investigation as part of the preoperative assessment, which also includes MRI of the rectum, ultrasound of the liver and chest X-ray (or abdominal /chest CT) to locate possible metastasis or synchronous tumors. However, it is often difficult to implement the preoperative colonic investigation due to lack of capacity or tumor stenosis. A recent Danish study showed that up to 78% of all patients with colorectal cancer had not received the full colonic investigation preoperatively. In this instance the recommendation from DCCG & DKS is that patients in the absence of complete colonic investigation preoperatively, should undergo colonoscopy within 3 months postoperatively.

Within the last 15 years new non-invasive imaging techniques have been developed, this includes MR colonography (MRC). Like conventional colonoscopy, MRC requires bowel cleansing, since feces can create artifacts that can hide or mimic polyps and abnormalities. After cleansing the colon is distended by water using a rectal catheter. Since it is only water that needs to pass through a possibly stenotic colon segment, there is a better chance to successfully examine the entire colon compared to a colonoscopy. A recent study showed a 98% success rate using MRC to examine the entire colon in patients with CRC having colon stenosis. The MRC is preformed after the colon is fully distended with water and depending on the resolution needed the scan times are between 10 and 15 minutes. Data processing, reconstruction and analysis are made at an independent workstation.

The advantages of MRC are its non-invasive nature, short examination time, and the fact that sedation is unnecessary. This makes it possible for patients to be discharged directly after the imaging procedure as opposed to the necessity for admission after a colonoscopy until the effects of the sedative drugs have worn off. Furthermore, it is assumed that patient compliance is much higher in MRC, since almost every patient finds it less unpleasant than colonoscopy.

MRI of the liver is a well-known procedure that has shown good results in the diagnosis of hepatic metastases and primary cancers. Several studies have shown that it is equal or better than CT and ultrasound of the liver.

Currently there are no studies, which make the overall preoperative assessment by means of one investigating technique, namely MRI. The investigators have previously studied the sensitivity/specificity and patient satisfaction by MRI colonography with fecal tagging. In this study the investigators want to investigate the quality of MR-colonography with bowel cleansing, also assessing the economical aspects of an overall examination of the rectum, colon and liver in patients with rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for operation for rectal cancer

Exclusion Criteria:

* Inflammatory bowel disease (IBD)
* Pacemaker
* Metal in the investigated areas
* Claustrophobia
* Age < 18 years
* Pregnancy
* Kidney disease
* Arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2010-08; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Synchronous colon cancers and liver metastasis | 2013 (up to 4 years)

SECONDARY OUTCOMES:
sensitivity/specificity of CT versus MR versus Peroperative ultrasonography of the liver | 2013 (up to 4 years)

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Achiam, MD, Ph.D., Principal Investigator — Herlev Hospital
Locations (1):
- Department of surgical gastroenterology, Copenhagen University Hospital at Herlev, Copenhagen, Denmark